CLINICAL TRIAL: NCT03964233
Title: A Phase Ia/Ib, Open Label, Dose-escalation Study of the Combination of BI 907828 (Brigimadlin) With BI 754091 (Ezabenlimab) and BI 754111 and the Combination of BI 907828 (Brigimadlin) With BI 754091(Ezabenlimab) Followed by Expansion Cohorts, in Patients With Advanced Solid Tumors
Brief Title: A Study in Patients With Different Types of Advanced Cancer (Solid Tumors) to Test Different Doses of BI 907828 (Brigimadlin) in Combination With BI 754091 (Ezabenlimab) and BI 754111 or BI 907828 (Brigimadlin) in Combination With BI 754091 (Ezabenlimab)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0002; 2019-001173-84 (EudraCT Number)
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — brigimadlin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation - BI 907828 + ezabenlimab (Experimental): All neoplasms
  Interventions: Drug: BI 907828; Drug: ezabenlimab
- Dose Expansion - Cohort 1 BI 907828 + ezabenlimab (Experimental)
  Interventions: Drug: BI 907828; Drug: ezabenlimab
- Dose Expansion - Cohort 2 - BI 907828 + ezabenlimab (Experimental)
  Interventions: Drug: BI 907828; Drug: ezabenlimab
- Dose Escalation - BI 907828 + ezabenlimab + BI 754111 (Experimental): All neoplasms
  Interventions: Drug: BI 907828; Drug: ezabenlimab; Drug: BI 754111

INTERVENTIONS:
Drug: BI 907828 — Film-coated tablets
  Other Names: Brigimadlin
Drug: ezabenlimab — Solution for infusion
  Other Names: BI 754091
Drug: BI 754111 — Solution for infusion
  Arms: Dose Escalation - BI 907828 + ezabenlimab + BI 754111

SUMMARY:
This study has 2 parts. The first part of the study is done. The first part was open to adults with different types of advanced cancer (solid tumors). The second part is open to people with specific types of soft tissue sarcoma, advanced lung cancer, and cancer in the stomach, bladder or bile ducts.

The participants get a combination of 2 medicines called brigimadlin (also called BI 907828) and ezabenlimab (also called BI 754091). Brigimadlin is a so-called MDM2 inhibitor that is being developed to treat cancer. Ezabenlimab is an antibody that may help the immune system fight cancer (immune checkpoint inhibitor). When the study started, some participants got a third medicine called BI 754111 in addition. Treatment with BI 754111 was stopped because data from another study showed no additional effect of BI 754111.

The purpose of the first part of the study was to find out the highest dose of brigimadlin that the participants could tolerate in combination with ezabenlimab. This dose is used in the second part of the study.

The purpose of the second part is to see whether the combination of brigimadlin with ezabenlimab is able to make tumors shrink.

The participants are in the study as long as they benefit from treatment and can tolerate it.

Ezabenlimab treatment is limited to 2 years. During this time, they get infusions of ezabenlimab, and take tablets with brigimadlin every 3 weeks. The doctors check how many participants have health problems during the study. The doctors also monitor the size of the tumor.

ELIGIBILITY:
Inclusion Criteria:

All cohorts:

* Provision of signed and dated, written informed consent form ICF in accordance with International Council on Harmonization-Good Clinical Practice (ICH-GCP)and local legislation prior to any trial-specific procedures, sampling, or analyses.
* Male or female ≥18 years old at the time of signature of the ICF.
* ECOG performance status of 0 or 1.
* Life expectancy of at least 12 weeks after the start of the treatment according to the Investigator's judgement.
* Patients with radiologically documented disease progression or relapse during or after all standard of care treatments. Patients who are not eligible to receive standard of care treatments, and for whom no proven treatments exist, are eligible.
* Previous treatment with an anti-PD-1/PD-L1 mAb is allowed as long as the last administration of the anti-PD-1/PD-L1 mAb on the previous treatment occurred a minimum of 28 days prior to the first administration of study treatment.
* Patient must be willing to participate in the blood sampling for the Pharmacokinetics (PK), Pharmacodynamics (PD), biomarker, and PGx analyses.
* Adequate organ function defined as all of the following (all screening labs should be performed locally within 10 days of treatment initiation):

  * Hematological

    * Absolute neutrophil count - ≥1.5 x 10^9/L
    * Platelets - ≥100 x 10^9/L
    * Hemoglobin 0 ≥8.5 g/dL or ≥5.3 mmol/L or ≥ 85 g/L
  * Hepatic

    * Total bilirubin ≤ 1,5 times the upper limit of normal (ULN), (patients with Gilbert's syndrome, total bilirubin must be < 3 x ULN)
    * Aspartate Transaminase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x ULN OR ≤5 x ULN for patients with liver metastases
  * Renal

    --- Creatinine - ≤1.5 x ULN - Patients may enter if creatinine is >1.5 x ULN and estimated glomerular filtration rate (eGFR) >50 mL/min (assessed by Chronic Kidney Disease Epidemiology [CKDEPI] Collaboration equation); confirmation of eGFR is only required when creatinine is >1.5 X ULN
  * Coagulation --- International Normalised Ratio (INR) or Prothrombin Time (PT). Activated Partial Thromboplastin Time (aPTT) - ≤1.5 x institutional ULN. Patients taking low dose warfarin must have their INR followed closely and according to institutional guidelines
* Women of childbearing potential (WOCBP, defined as female patients who are premenopausal or who had no cessation of menses within 12 months without an alternative medical cause, but not including female patients who are permanently sterilized) and men able to father a child must be ready and able to use two medically acceptable methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at screening, during trial participation. A list of contraception methods meeting these criteria is provided in the patient information.

Phase Ia (dose escalation part):

* Patients with a confirmed diagnosis of unresectable, advanced and/or metastatic solid tumors (any type) irrespective of the TP53 mutation status,
* Patient with either evaluable or non-evaluable disease.
* Availability and willingness to provide a sample of archival Formalin-fixed paraffin embedded (FFPE) tumor tissue material

Phase Ia (Expansion Cohort):

* Patients with MDM2 amplified tumors and TP53 wild type status confirmed on tumor tissue
* At least one target lesion that can be accurately measured per RECIST 1.1. In patients who only have one target lesion, the baseline imaging must be performed at least two weeks after any biopsy of the target lesion.

Phase Ib (dose expansion part):

* At least one target lesion that can be accurately measured per RECIST 1.1. In patients who only have one target lesion, the baseline imaging must be performed at least two weeks after any biopsy of the target lesion.
* Patients with TP53 wild-type status confirmed on tumor tissue. Provision of fresh tissue biopsy at screening (may be omitted if patient has archival tissue within 12 months prior to enrolment) and willingness to provide fresh tissue biopsy on study, if safe and feasible on either occasion
* Expansion cohorts:

  * Cohort 1: Patients with unresectable, advanced and/or metastatic TP53 wt one line of systemic medical treatment in the advanced and/or metastatic setting: Liposarcoma excluding dedifferentiated liposarcoma, Undifferentiated pleomorphic sarcoma, Myxofibrosarcoma, Synovial sarcoma, Leiomyosarcoma
  * Cohort 2: Patients with unresectable, advanced and/or metastatic TP53 wt MDM2-amplified tumors as listed below, who received at least one line of systemic medical treatment in the advanced and/or metastatic setting: NSCLC (patients with NSCLC harboring genomic aberrations for which approved targeted therapy is approved and available, must have received such prior treatment), Gastric adenocarcinoma, Urothelial carcinoma, Biliary tract carcinoma (including cholangiocarcinoma, intra-and extrahepatic biliary tree, gall bladder and ampulla of vater)

Exclusion criteria:

* Previous administration of BI 907828 or any other MDM2-p53 or MDMX (MDM4)-p53 antagonist
* In Phase Ib (expansion phase) and Phase Ia expansion cohort only: a documented amino-acid altering mutation in TP53 occurring in the patient's tumor.
* Symptomatic brain metastases. Note: Patients with previously treated brain metastases may participate but treated lesions should not be used as target lesions
* Active bleeding, significant risk of haemorrhage (e.g. previous severe gastrointestinal bleeding, previous haemorrhagic stroke at any time), or current bleeding disorder (e.g. haemophilia, von Willebrand disease)
* Major surgery (major according to the Investigator's assessment) performed within 12 weeks prior to start of study treatment, or planned within 12 months after screening (e.g. hip replacement).
* Any other documented active or suspected malignancy or history of malignancy within 3 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Currently enrolled in another investigational device or drug trial, or less than 4 weeks since receiving other investigational treatments. Patients who are in follow-up/observation for another clinical trial are eligible.
* Patients who have not recovered from all clinically significant adverse events from their most recent therapy or intervention prior to study enrolment
* Known history of human immunodeficiency virus (HIV) infection
* Any of the following laboratory evidence of hepatitis virus infection:

  * Positive results of hepatitis B surface (HBs) antigen
  * Presence of HBc antibody together with HBV-DNA
  * Presence of hepatitis C RNA
* Known hypersensitivity to the trial drugs or their excipients.
* Serious concomitant disease or medical condition affecting compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the Investigator, would make the patient inappropriate for entry into the trial.
* Chronic alcohol or drug abuse or any condition that, in the Investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial; female patients who do not agree to the interruption of breast feeding from the start of study treatment to within 30 days after the last study treatment.
* History (including current) of interstitial lung disease or pneumonitis within the last 5 years.
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of study treatment.
* Active autoimmune disease or a documented history of autoimmune disease, disease, that requires systemic treatment, i.e. corticosteroids or immunosuppressive drugs, except vitiligo or resolved childhood asthma/atopyatopy, alopecia, or any chronic skin condition that does not require systemic therapy; patients with autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and/or controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible.
* Active infection requiring systemic treatment (antibacterial, antiviral, or antifungal therapy) at start of treatment in this trial.
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) >470 msec
  * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block
  * Any factor that increases the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval
  * Patients with an ejection fraction (EF) <50% or the lower limit of normal of the institutional standard will be excluded. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF, will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g., echocardiogram, multi-gated acquisition scan). A historic measurement of EF no older than 6 months prior to first administration of study drug can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or of the treating physician or both.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
Phase Ia - maximum tolerated dose (MTD) of brigimadlin (BI 907828) in combination with ezabenlimab based on the number of patients with dose limiting toxicities (DLTs) during the first treatment cycle | Up to 21 Days
Phase Ib - Objective response (OR) | Up to 24 months
Phase Ib - Progression free survival | Up to 24 months

SECONDARY OUTCOMES:
Phase Ia - Cmax : Maximum measured plasma concentration of brigimadlin (BI 907828) and ezabenlimab (during the first cycle) | Up to 21 Days
Phase Ia - AUC0-tz: Area under the concentration-time curve in plasma for brigimadlin (BI 907828) and ezabenlimab over the time interval from 0 to the last quantifiable time point (during the first cycle) | Up to 21 Days
Phase Ia - Number of patients with DLTs observed during the entire treatment period | Up to 24 months
Phase Ib - Objective Response (OR) | Up to 24 months
Phase Ib - Disease control (DC) | Up to 24 months
Phase Ib - Number of patients with DLTs | Up to 2 years
Phase Ib - Overall survival (OS) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (23):
- United States (9):
  - Sarcoma Oncology Center, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - University Cancer and Blood Center, Athens, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology-Irving-69444, Irving, Texas
  - NEXT Oncology-San Antonio-65273, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- Linear Clinical Research, Nedlands, Western Australia, Australia
- UZ Leuven, Leuven, Belgium
- France (3):
  - INS Bergonie, Bordeaux
  - CTR Leon Berard, Lyon
  - INS Gustave Roussy, Villejuif
- Germany (2):
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Ulm, Ulm
- Central Hospital of Northern Pest - Military Hospital, Budapest, Hungary
- National Cancer Center Hospital, Tokyo, Chuo-ku, Japan
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- National Cancer Centre Singapore, Singapore, Singapore
- Spain (2):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid
- The Royal Marsden Hospital, Chelsea, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency